CLINICAL TRIAL: NCT06270394
Title: Fibroblast Activation Protein PET/CT or PET/MR Production in the Diagnosis, Staging, and Efficacy Assessment of Malignant Tumors Application
Brief Title: FAP PET/CT or PET/MR Production in the Diagnosis, Staging, and Efficacy Assessment of Malignant Tumors Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MJX
Record Dates: First submitted 2024-01-23; First posted 2024-02-21 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Malignant Tumors; Positron-Emission Tomography
Keywords: FAPI; PET/CT; PET/MRI; Malignant Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI PET/MRI scan (Experimental): The 68Ge/68Ga generator was eluted with 0.1 M HCL solution to achieve 3.0 ml of liquid, which was mixed thoroughly with 20 µg FAPI precursor and 375 µl of 1.25 M sodium acetate. The mixture was placed in a thermostat at 95°C for 10 min. The finished liquid was passed through an activated Sep-pak 18C column and 0.8 ml of 80% ethanol was passed through the Sep-pak 18C column and a 0.2 µm microporous membrane (Pall Co., Ltd.) before the product was collected in a sterile product vial.
  The equipment scan pf PET/MRI is the SIGNA PET/MR manufactured by GE Healthcare. The scan is performed approximately 40 min after injection of 1.85-3.7 MBq 68Ga-FAPI-04 per kg body weight. Breath-gated corrected step-and-shoot (SS) acquisition mode was used. The scan time was 60 ± 10 min (50-70 min). Dedicated T1- and T2-weighted images and diffusion-weighted images (DWI) of the head and neck, chest, abdomen, and pelvis were acquired.
  Interventions: Drug: 68Ga-Fibroblast activation protein inhibitor

INTERVENTIONS:
Drug: 68Ga-Fibroblast activation protein inhibitor — Fibroblast activation protein (FAP), a type II transmembrane serine protease with dipeptidyl peptidase and endopeptidase activities. FAP is a specific surface marker for activated fibroblasts in the mesenchyme of tumors, which account for 90% of the stroma of epithelial neoplasms. FAP inhibitors (FAPIs) can specifically target and bind to FAP. These inhibitors that are radiolabeled with gallium 68 (68Ga-FAPIs) can be probes for visualization of the FAP tumor stroma. Previous studies have demonstrated that 68Ga-FAPI-04 is not dependent on blood glucose levels, has an equal or better tumor-to-background ratio, and clearly visualizes primary tumors and their metastatic foci. In addition, previous studies on 68Ga-FAPI-04 have focused on PET/CT and the efficacy of PET/MR with FAPI for postoperative evaluation of GI tumors remains to be clarified.
  Other Names: PET-MRI (SIGNA PET/MR manufactured by GE Healthcare)

SUMMARY:
This clinical trial aims to investigate the value of fibroblast activation protein PET/CT(PET/MR) in the diagnosis, staging, and evaluation of treatment outcomes in malignant tumors. The main question it aims to answer is:

Fibroblast Activation Protein PET/CT(PET/MR) whether or in which cases this assay is superior to conventional FDG examination in the diagnosis, staging, and assessment of therapeutic efficacy of malignant tumors, thinking about the reasons behind this.

Investigators will screen suitable participants among patients undergoing routine FDG examination.

* Participants will sign an informed consent form
* Undergo 68Ga-FAPI PET/CT (PET/MR) before surgery or biopsy
* Surgical resection or puncture biopsy to obtain pathologic results. Diagnosis of patients with malignant tumors at first diagnosis; clinical staging of tumors; and clinical outcomes of patients with confirmed diagnoses will be assessed after postoperative investigator follow-up.

The researchers will compare the FDG exams the participants have had to determine the effectiveness of the fibroblast activating protein test.

DETAILED DESCRIPTION:
1. Title of research program Fibroblast activation protein(AFP) Positron Emission Tomography(PET)-CT or -MR production in the diagnosis of malignant tumors, staging and therapeutic evaluation of clinical applications.

   Application.
2. Background Currently, 18F-FDG PET is one of the most commonly used methods for diagnosis, staging, efficacy assessment, and prognosis evaluation of malignant tumors. The basic principle of 18F-FDG PET is the Warburg effect. However, 18F-FDG has its limitations, such as low specificity, low detection rate of small tumors, mucin-secreting epithelial malignant tumors, squamous cell carcinomas, highly differentiated neuroendocrine tumors, squamous cell carcinomas, highly differentiated neuroendocrine tumors, and highly differentiated endocrine gland malignancies, among others, have low uptake.

18F-FDG is a non-specific metabolic PET tracer that can reflect glucose metabolism in malignant tumors. However, 18F-FDG can also be taken up by inflammatory lesions, infectious lesions, benign tumors, etc. Therefore, 18F-FDG tumor imaging has relative limitations. Nowadays, molecular imaging is changing from non-specific to specific radiotracer imaging. Therefore, tumor-associated fibroblasts (CAFs) have gradually become a new research hotspot.

Fibroblasts are the main host cells in the tumor microenvironment and are also the main stromal cells of solid tumors, they can interact with tumor cells, make their own morphology and physiological function changes, express a variety of cytokines, proteases, adhesion, molecular, different degree increase of tumor cell malignant characterization, and the occurrence of tumor, growth, blood vessel formation, invasion is closely related to metastasis. It has been confirmed that FAP is expressed in melanoma, colorectal cancer, breast cancer, pancreatic cancer, gastric cancer, lung cancer, esophageal cancer, ovarian cancer, cervical cancer, endometrial cancer, oral squamous cell carcinoma, and osteosarcoma, etc., and is associated with tumor growth and invasion. FAPαis a type II transmembrane glycoprotein, consisting of a primary chain of 760 amino acids with a small intracellular component or short cytoplasmic tail (6 amino acids), a transmembrane component (19 amino acids) and a large extracellular component. The monomeric form of FAPα is inactive but is activated by polymerization activity through polymerization-activation to form either the homodimer FAPα/FAPα or the heterodimer FAPα/FAPβ. This membrane-bound protein is one of the key components of the extracellular matrix and plays an important role in regulating or remodeling the tumor microenvironment. Fibroblast activation protein inhibitor Preparation (FAPI) is a novel class of probes, and the enzymatic activity of FAP provides a new diagnostic and therapeutic target. Therefore, the selection of FAPI to target FAP overexpression induced by tumor-associated fibroblasts has become a new research hotspot. Currently, new molecules such as FAPI-02, FAPI-04, FAPI-46, and other inhibitory ligands have been designed, synthesized, and conducted in vitro and in vivo experiments. Because the biological half-life of these probes matches the physical half-life of gallium-68 (Ga-68), if these molecules form new molecules after being labeled with Ga-68, the new molecules become very promising molecular probes for research. PET/CT has been gradually applied to the examination of malignant tumors, and can be used for the diagnosis of tumors, clinical staging, and evaluation of therapeutic efficacy. PET/MRI is an emerging molecular imaging method in recent years. With the popularization of integrated PET/MR imaging, combining the higher resolution and morphology of MR imaging with the N-staging and M-staging of PET has greatly improved the detection rate of some tumors and the degree of tissue invasion around the lesion. In this study, investigators propose to use fibroblast activation protein PET/CT and PET/MR for the diagnosis, staging, and evaluation of treatment effects of malignant tumors, to evaluate its real value and to make up for the insufficiency of 18F-FDG PET/CT.

3. Research objectives To study the value of FAPI PET/CT and PET/MR in diagnosing, staging, and evaluating treatment effects of malignant tumors.

4. Types of study design, method of randomization, and level of blinding Type of study design: observational study (prospective study).

5. Criteria for selection of participants

* 18 years ≤ 75 years of age;
* Patients with clinical suspicion of malignancy;
* No invasive tests or treatments recently;
* Blood routine: leukocyte > 4×10 9/L, neutrophil > 2×10 9/L, hemoglobin > 90g/L, platelets > 100×10 9/L;
* Cardiac function: left ventricular ejection fraction >50%;
* Pulmonary function tests: FEV1 ≥1.2L, FEV1% ≥50% and DLCO ≥50%;
* Liver function: total bilirubin <1.5 times upper limit of normal (ULN); AST and ALT <1.5 times ULN;
* Renal function: serum creatinine ≤ 1.5 times ULN, or glomerular filtration rate > 60 ml/min;
* Participants agreed to participate in this clinical trial and signed an informed consent form;
* Good compliance and commitment to follow the study procedures and to cooperate in the implementation of the full study;
* No birth plans for six months.

  6. Exclusion criteria for participants
* Those with severe psychiatric symptoms, or those who are too confused to cooperate with the examination;
* Pregnant and potentially pregnant women, lactating women;
* Those with poor compliance.

  7. Calculate based on statistical principles, the number of cases required to achieve the desired purpose of the study This was an exploratory observational study and the sample size was not calculated based on statistical assumptions, and the sample size was initially determined to be 60 cases.

  8. Technology road map

  9. Criteria for discontinuing clinical studies, provisions for ending clinical studies
  1. Significant errors in the clinical research protocol or serious deviations in the implementation of the protocol that make it difficult to assess the utility of the study;
  2. The drug regulatory authority, government department or ethics committee asked to suspend or end the study;
  3. Circumstances in which other researchers do not consider it appropriate to continue the study or find it difficult to do so.

  10. Participant screening number, participant number, and case report form are maintained participant Screening Number: a 1-sequential number, e.g., 1-1 for the first participant; participant Number: a sequential number, e.g., 001 for the first participant; Case report form retention: information is entered into the CRF form by the project leader or other authorized investigator, and only medically qualified investigators are allowed to complete the original clinical assessment/safety data. Any changes made to the CRF form by the project leader or other authorized researchers after the original data has been entered need to be documented. Any modification of data that has been endorsed will require the name of the researcher or other authorized researcher who modified it, the date of the modification, and the reason for the modification (if the change is minor).

  11. Documentation of adverse events and methods of reporting serious adverse events, management measures, modalities, timing and fate of follow-up visits 11.1Adverse events Adverse Event (AE) is an unfavorable medical event that occurs during a clinical trial. Clinical trial Any adverse event that occurs during the implementation should be faithfully recorded and analyzed for reasons. Both anticipated and unanticipated adverse events should be recorded and reported truthfully. Adverse events should be included as outcome variables in the statistical analysis of clinical trials.

11.2Serious adverse event A serious Adverse Event (SAE) is a clinical trial event that results in death or serious deterioration of health, including fatal illness or injury, permanent defects in body structure or function, hospitalization or prolonged hospitalization, or the need for medical or surgical intervention to avoid permanent defects in body structure or function. Events that result in fetal distress, fetal death, or congenital anomalies or congenital defects.

11.3Reporting procedures 11.3.1Reporting time frames In the event of AE or SAE in this clinical trial, the investigator shall immediately take appropriate therapeutic measures for the participant, notify the principal investigator, and report in writing to the appropriate authorities within 24 hours once SAE has been determined.

11.3.2Reporting Sector The office of the clinical trial organization to which it belongs, the sponsor, our Ethics Committee, as well as the drug supervision and management department of the province, autonomous region, and municipality directly under the central government where the clinical trial organization is located, and the competent department of health and wellness.

11.3.3Reporting methods If an SAE occurs, the investigator completes the Adverse Event Record Form and files the original Adverse Event Record Form in the investigator's file folder.

11.3.4Processing and recording When an SAE or suspected SAE occurs, the investigator immediately stops the trial and takes appropriate therapeutic measures, notifies the principal investigator and the sponsor; the principal investigator makes a judgment about the relevance of the SAE to the trial and records the occurrence, development, and treatment of the SAE in as much detail as possible on the Adverse Event Record Form, which is documented on the Case Report Form, signed and dated.

11.3.5follow-up If SAE is determined, the event must be followed until it appears to improve, stabilizes, or, in the judgment of the principal investigator, does not require follow-up.

12. Statistical analysis plan, definition, and selection of data sets for statistical analysis 12.1General approach SPSS software was used for statistical analysis of data. If the data were normally distributed, they were expressed as mean ± standard deviation and compared using a two-sample t-test and one-way ANOVA. If the data were not normally distributed, they were expressed as M(P5, P95) and compared using the Mann-Whitneyu and Kruskal-WallisH rank sum tests. P<0.05 is considered a statistically significant difference.

12.2Analysis of Primary and Secondary Study Endpoints Survival analysis was performed using the Kaplan-Meier method to plot survival curves, and the log-rank test was used to compare survival differences between groups.

13. Data management and confidentiality of information 13.1Data entry and modification Data entry and modification will be done by the Department of Nuclear Medicine, and data collection will be performed by clinical researchers under the supervision of the person in charge, who will be responsible for the accuracy, completeness, and timeliness of the reported data. All data should be clear to ensure accurate interpretation and traceability. Clinical data will be maintained in a database, which should be password-protected, and a logical proofreading process should be in place when the database is created.

The Data Manager is responsible for reviewing and managing the entered data. In case of doubt about the existence of data, the data manager will send the appropriate query to the researcher, who will respond to the query sent by the data manager promptly, and the data manager will be able to re-question the data if necessary.

13.2Confidentiality Program for Research Participant Information Participant's personal information follows the principle of confidentiality. The investigator will replace the participants' identifying information with a code name that does not contain participants' name.

13.3Confidentiality Program for Research Data

14. Quality control and quality assurance in clinical research 14.1Conditions of research units and training of personnel The department in which the research project is located has the appropriate personnel, equipment, and first aid facilities; All research participants (including doctors, nurses, and others) have received appropriate training about the research and any information relevant to the conduct of the research has been passed on to the relevant personnel; All equipment has a technical inspection certificate from the technical supervision department indicating that it is in good working order; During the trial study, the investigators should be relatively fixed, and for the change of investigators in the middle of the study, they should join the study after training, and the "Clinical Trial Participant Contact Form" should be changed again.

14.2Modifications to the pilot program Any modifications to the trial protocol that would affect the execution of the study, the purpose of the trial, the design of the trial, the number of patient cases and the flow of the trial, etc., must be submitted as amendments to the trial protocol, which must be agreed upon by the investigator and the Ethics Committee before they can be implemented.

15. Study of related ethics Participants are not paid and do not incur any costs. The study was conducted by China's Measures for Ethical Review of Biomedical Research Involving Human Beings and international ethical guidelines such as the Declaration of Helsinki.

16. Participant recruitment methods and the process of obtaining informed consent Participant Recruitment Methods: Patients meeting the inclusion/exclusion criteria were referred by the Department of Nuclear Medicine for inclusion in the clinical study.

Informed Consent Process: Informed consent should be completed before the participant agrees to participate in the study and should continue throughout the study. The informed consent form was agreed upon by the Ethics Committee and should be read and signed by the participants. The researcher will explain the research process answer questions from participants and inform participants of the possible risks and their rights. Participants may discuss with a family member or guardian before agreeing to participate. The investigator must inform participants that participation in the study is voluntary and that they may withdraw from the study at any time during the study. A copy of the informed consent form can be provided to the study participant to keep. The rights and welfare of subjects will be protected and it is emphasized that the quality of their medical care will not be compromised by refusal to participate in research.

17. Expected progress and completion date of the clinical study 2022.4.28-2027.3.31 Screening of eligible participants, who underwent relevant examinations as arranged by the investigator; 2027.4.1-2027.9.30 Complete the statistical analysis of the experimental data.

18. Follow-up and medical measures at the end of the study Patients are followed up on a long-term basis and assistance is provided accordingly.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ 75 years of age;
* Patients with clinical suspicion of malignancy;
* No invasive tests or treatments recently;
* Blood routine: leukocyte > 4×109/L, neutrophil > 2×10 9/L, hemoglobin > 90g/L, platelets > 100×10 9/L;
* Cardiac function: left ventricular ejection fraction >50%;
* Pulmonary function tests: FEV1 ≥1.2L, FEV1% ≥50% and DLCO ≥50%;
* Liver function: total bilirubin <1.5 times upper limit of normal (ULN); AST and ALT <1.5 times ULN;
* Renal function: serum creatinine ≤ 1.5 times ULN, or glomerular filtration rate > 60 ml/min;
* Participants agreed to participate in this clinical trial and signed an informed consent form;
* Good compliance and commitment to follow the study procedures and to cooperate in the implementation of the full study;
* No birth plans for six months.

Exclusion Criteria:

* Those with severe psychiatric symptoms, or those who are too confused to cooperate with the examination;
* Pregnant and potentially pregnant women, lactating women;
* Those with poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
68Ga-Fibroblast Activation Protein Inhibitor-04 Uptake in Gastrointestinal Cancer: Comparison with 18F-FDG | up to 38 months
  18F-FDG PET/CT and 68Ga-FAPI-04 PET/MR scans were acquired independently for all the participants with pathologically confirmed GI tumors and signs. The χ2 test was used to analyze these two technologies to quantitatively compare the diagnostic effects. The normalized SUVmax values (calculated by dividing a lesion's original SUVmax by the SUVmean of the descending aorta) of selected lesions were measured and analyzed by Student's t-test. A visual assessment system of the regions was prepared.

SECONDARY OUTCOMES:
Utility of 68Ga-FAPI-04 PET/MRI combines 18F-FDG PET/CT in the postoperative evaluation of gastrointestinal cancers | up to 60 months
  18F-FDG PET/CT and 68Ga-FAPI-04 PET/MR scans were acquired independently for all the participants with pathologically confirmed GI tumors and signs. The χ2 test was used to analyze these two technologies to quantitatively compare the diagnostic effects. The normalized SUVmax values (calculated by dividing a lesion's original SUVmax by the SUVmean of the descending aorta) of selected lesions were measured and analyzed by Student's t-test. A visual assessment system of the regions was prepared. A visual scoring system was established to compare the detectability of primary tumors and metastases in different organs or regions (the peritoneum, abdominal lymph nodes, supradiaphragmatic lymph nodes, liver, ovary, bone, and other tissues).

CONTACTS AND LOCATIONS:
Overall Officials: Huiqin Xu, Study Chair — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- FirstHAnhuiMU, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the current study are available from the Study Chair upon reasonable request.

REFERENCES:
- [Background] Warburg O, Wind F, Negelein E. THE METABOLISM OF TUMORS IN THE BODY. J Gen Physiol. 1927 Mar 7;8(6):519-30. doi: 10.1085/jgp.8.6.519. No abstract available. PMID 19872213
- [Background] Mankoff DA, Eary JF, Link JM, Muzi M, Rajendran JG, Spence AM, Krohn KA. Tumor-specific positron emission tomography imaging in patients: [18F] fluorodeoxyglucose and beyond. Clin Cancer Res. 2007 Jun 15;13(12):3460-9. doi: 10.1158/1078-0432.CCR-07-0074. PMID 17575208
- [Background] Chang JM, Lee HJ, Goo JM, Lee HY, Lee JJ, Chung JK, Im JG. False positive and false negative FDG-PET scans in various thoracic diseases. Korean J Radiol. 2006 Jan-Mar;7(1):57-69. doi: 10.3348/kjr.2006.7.1.57. PMID 16549957
- [Background] Cheng JD, Valianou M, Canutescu AA, Jaffe EK, Lee HO, Wang H, Lai JH, Bachovchin WW, Weiner LM. Abrogation of fibroblast activation protein enzymatic activity attenuates tumor growth. Mol Cancer Ther. 2005 Mar;4(3):351-60. doi: 10.1158/1535-7163.MCT-04-0269. PMID 15767544
- [Background] Pineiro-Sanchez ML, Goldstein LA, Dodt J, Howard L, Yeh Y, Tran H, Argraves WS, Chen WT. Identification of the 170-kDa melanoma membrane-bound gelatinase (seprase) as a serine integral membrane protease. J Biol Chem. 1997 Mar 21;272(12):7595-601. doi: 10.1074/jbc.272.12.7595. PMID 9065413
- [Background] Huber MA, Kraut N, Park JE, Schubert RD, Rettig WJ, Peter RU, Garin-Chesa P. Fibroblast activation protein: differential expression and serine protease activity in reactive stromal fibroblasts of melanocytic skin tumors. J Invest Dermatol. 2003 Feb;120(2):182-8. doi: 10.1046/j.1523-1747.2003.12035.x. PMID 12542520
- [Background] Henry LR, Lee HO, Lee JS, Klein-Szanto A, Watts P, Ross EA, Chen WT, Cheng JD. Clinical implications of fibroblast activation protein in patients with colon cancer. Clin Cancer Res. 2007 Mar 15;13(6):1736-41. doi: 10.1158/1078-0432.CCR-06-1746. PMID 17363526
- [Background] Shi M, Yu DH, Chen Y, Zhao CY, Zhang J, Liu QH, Ni CR, Zhu MH. Expression of fibroblast activation protein in human pancreatic adenocarcinoma and its clinicopathological significance. World J Gastroenterol. 2012 Feb 28;18(8):840-6. doi: 10.3748/wjg.v18.i8.840. PMID 22371645
- [Background] Goscinski MA, Suo Z, Florenes VA, Vlatkovic L, Nesland JM, Giercksky KE. FAP-alpha and uPA show different expression patterns in premalignant and malignant esophageal lesions. Ultrastruct Pathol. 2008 May-Jun;32(3):89-96. doi: 10.1080/01913120802034934. PMID 18570153
- [Background] Lai D, Ma L, Wang F. Fibroblast activation protein regulates tumor-associated fibroblasts and epithelial ovarian cancer cells. Int J Oncol. 2012 Aug;41(2):541-50. doi: 10.3892/ijo.2012.1475. Epub 2012 May 14. PMID 22614695
- [Background] Rasanen K, Virtanen I, Salmenpera P, Grenman R, Vaheri A. Differences in the nemosis response of normal and cancer-associated fibroblasts from patients with oral squamous cell carcinoma. PLoS One. 2009 Sep 1;4(9):e6879. doi: 10.1371/journal.pone.0006879. PMID 19721715
- [Background] Dohi O, Ohtani H, Hatori M, Sato E, Hosaka M, Nagura H, Itoi E, Kokubun S. Histogenesis-specific expression of fibroblast activation protein and dipeptidylpeptidase-IV in human bone and soft tissue tumours. Histopathology. 2009 Oct;55(4):432-40. doi: 10.1111/j.1365-2559.2009.03399.x. PMID 19817894
- [Background] Cheng JD, Dunbrack RL Jr, Valianou M, Rogatko A, Alpaugh RK, Weiner LM. Promotion of tumor growth by murine fibroblast activation protein, a serine protease, in an animal model. Cancer Res. 2002 Aug 15;62(16):4767-72. PMID 12183436
- [Background] Liu R, Li H, Liu L, Yu J, Ren X. Fibroblast activation protein: A potential therapeutic target in cancer. Cancer Biol Ther. 2012 Feb 1;13(3):123-9. doi: 10.4161/cbt.13.3.18696. Epub 2012 Feb 1. PMID 22236832
- [Background] Giesel FL, Kratochwil C, Lindner T, Marschalek MM, Loktev A, Lehnert W, Debus J, Jager D, Flechsig P, Altmann A, Mier W, Haberkorn U. 68Ga-FAPI PET/CT: Biodistribution and Preliminary Dosimetry Estimate of 2 DOTA-Containing FAP-Targeting Agents in Patients with Various Cancers. J Nucl Med. 2019 Mar;60(3):386-392. doi: 10.2967/jnumed.118.215913. Epub 2018 Aug 2. PMID 30072500
- [Background] Hathi DK, Jones EF. 68Ga FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. Radiol Imaging Cancer. 2019 Sep 27;1(1):e194003. doi: 10.1148/rycan.2019194003. eCollection 2019 Sep. No abstract available. PMID 33778675
- [Background] Loktev A, Lindner T, Burger EM, Altmann A, Giesel F, Kratochwil C, Debus J, Marme F, Jager D, Mier W, Haberkorn U. Development of Fibroblast Activation Protein-Targeted Radiotracers with Improved Tumor Retention. J Nucl Med. 2019 Oct;60(10):1421-1429. doi: 10.2967/jnumed.118.224469. Epub 2019 Mar 8. PMID 30850501
- See also: THE METABOLISM OF TUMORS IN THE BODY — https://pubmed.ncbi.nlm.nih.gov/19872213/
- See also: Tumor-specific positron emission tomography imaging in patients: [18F] fluorodeoxyglucose and beyond — https://pubmed.ncbi.nlm.nih.gov/17575208/
- See also: False positive and false negative FDG-PET scans in various thoracic diseases — https://pubmed.ncbi.nlm.nih.gov/16549957/
- See also: Abrogation of fibroblast activation protein enzymatic activity attenuates tumor growth — https://pubmed.ncbi.nlm.nih.gov/15767544/
- See also: Identification of the 170-kDa melanoma membrane-bound gelatinase (seprase) as a serine integral membrane protease — https://pubmed.ncbi.nlm.nih.gov/9065413/
- See also: Fibroblast activation protein: differential expression and serine protease activity in reactive stromal fibroblasts of melanocytic skin tumors — https://pubmed.ncbi.nlm.nih.gov/12542520/
- See also: Clinical implications of fibroblast activation protein in patients with colon cancer — https://pubmed.ncbi.nlm.nih.gov/17363526/
- See also: Expression and role of fibroblast activation protein-alpha in micro-invasive breast carcinoma — https://pubmed.ncbi.nlm.nih.gov/22067528/
- See also: Expression of fibroblast activation protein in human pancreatic adenocarcinoma and its clinicopathological significance — https://pubmed.ncbi.nlm.nih.gov/22371645/
- See also: FAP-alpha and uPA show different expression patterns in premalignant and malignant esophageal lesions — https://pubmed.ncbi.nlm.nih.gov/18570153/
- See also: Fibroblast activation protein regulates tumor-associated fibroblasts and epithelial ovarian cancer cells — https://pubmed.ncbi.nlm.nih.gov/22614695/
- See also: Differences in the nemosis response of normal and cancer-associated fibroblasts from patients with oral squamous cell carcinoma — https://pubmed.ncbi.nlm.nih.gov/19721715/
- See also: Histogenesis-specific expression of fibroblast activation protein and dipeptidylpeptidase-IV in human bone and soft tissue tumours — https://pubmed.ncbi.nlm.nih.gov/19817894/
- See also: Promotion of tumor growth by murine fibroblast activation protein, a serine protease, in an animal model — https://pubmed.ncbi.nlm.nih.gov/12183436/
- See also: Fibroblast activation protein: A potential therapeutic target in cancer — https://pubmed.ncbi.nlm.nih.gov/22236832/
- See also: 68Ga-FAPI PET/CT: Biodistribution and Preliminary Dosimetry Estimate of 2 DOTA-Containing FAP-Targeting Agents in Patients with Various Cancers — https://pubmed.ncbi.nlm.nih.gov/30072500/
- See also: 68Ga FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer — https://pubmed.ncbi.nlm.nih.gov/33778675/
- See also: Radiation dosimetry and biodistribution of 68Ga-FAPI-46 PET imaging in cancer patients — https://pubmed.ncbi.nlm.nih.gov/31836685/
- See also: Development of Fibroblast Activation Protein-Targeted Radiotracers with Improved Tumor Retention — https://pubmed.ncbi.nlm.nih.gov/30850501/